CLINICAL TRIAL: NCT03358537
Title: A Low-residue Diet is a Good Option for Patients With PEG Based Colon Preparation: a Randomized Clinical Trial
Brief Title: A Low-residue Diet vs Clear Liquid Diet as a Bowel Colonoscopy Preparation With Polyethylene Glycol (PEG)
Acronym: PEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, FELIX IGNACIO TELLEZ AVILA, M.D., M.Sc., Ph. D, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 001157
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Colonoscopy
Keywords: Dietary fiber

STUDY DESIGN:
Intervention Model Description: A total of 215 subjects were randomly assigned for this study, 105 in the clear liquid diet and 100 in the low residue-diet, 5 subjects were excluded in each group
Who Masked: Care Provider
Masking Description: This was a randomized, endoscopists' blinded comparison of bowel cleanising, tolerability and quality indicators for colonoscopy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clear Liquid Diet (Active Comparator): 110 subjects received clear liquid diet 24 hours before colonoscopy
  Interventions: Dietary Supplement: Clear Liquid Diet
- Low-residue Diet (Active Comparator): 105 subjects received a prespecified low-residue diet 24 hours before colonoscopy
  Interventions: Dietary Supplement: Low-residue Diet

INTERVENTIONS:
Dietary Supplement: Clear Liquid Diet — Clear liquid diet was compared with low-residue diet, in combination with Poliethylene Glycol in each group
  Arms: Clear Liquid Diet
Dietary Supplement: Low-residue Diet — Clear liquid diet was compared with low-residue diet, in combination with Poliethylene Glycol in each group
  Arms: Low-residue Diet

SUMMARY:
This was a randomized, endoscopists' blinded comparison of bowel colonoscopy cleansing and tolerability of a prespecified low-residue diet compared with a clear liquid diet and Polyethylene Glycol bowel preparation. Outcome measures included efficacy of bowel preparation, patient preparation tolerability and side-effects.

DETAILED DESCRIPTION:
An adequate examination is dependent on the bowel colonoscopy cleansing of stool. There are many different colon preparations, however endoscopists traditionally recommend the patient remain on a clear liquid diet for at least 24 h prior to their colonoscopy to reduce continued residue inflow into the colon from the small bowel, in addition the large volume preparation with PEG. The most common problems leading to less than adequate colon cleansing include lack of compliance with the clear liquid diet and difficulty taking the large volume preparation.

ELIGIBILITY:
Inclusion Criteria:

* Out-patient scheduled for colonoscopy

Exclusion Criteria:

* Subjects under 18 years of age
* Pregnancy
* Subjects with decompensated metabolic, renal, cardiac and psychiatric disease
* Allergy to PEG
* Refuse participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Quality of bowel colonoscopy preparation | 1 day
  The quality of cleansing was recorded using the Boston Bowel Preparation Scale (BBPS), a four-point scoring system applied to each of the three broad regions of the colon (right=cecum and ascending, transverse= including the hepatic and splenic flexures and left=descending, sigmoid and rectum) during withdrawal. The point was assigned as 0= unprepared to 3=entire mucosa of colon segment seen well with no residual staining. Successful colon cleansing was considered when BBPS were >2 per segment.

SECONDARY OUTCOMES:
Tolerability | 1 day
  Patient tolerability was assessed using Viera scale (Likert), which measures the intensity of the symptoms related to the bowel preparation including nausea, vomiting, abdominal pain, abdominal distension and anal discomfort. The six-point scale ranging from 0-1=no complaints or some; 2-3=moderate and 4-5=severe symptoms.
Satisfaction | 1 day
  Data on satisfaction were collected with a 1 to 10 visual analogue scale. Volume PEG consumed were evaluated as quartile (0%, 25%, 50%, 75% and 100%) prior colonoscopy.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delegge M, Kaplan R. Efficacy of bowel preparation with the use of a prepackaged, low fibre diet with a low sodium, magnesium citrate cathartic vs. a clear liquid diet with a standard sodium phosphate cathartic. Aliment Pharmacol Ther. 2005 Jun 15;21(12):1491-5. doi: 10.1111/j.1365-2036.2005.02494.x. PMID 15948817
- [Result] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Result] Park DI, Park SH, Lee SK, Baek YH, Han DS, Eun CS, Kim WH, Byeon JS, Yang SK. Efficacy of prepackaged, low residual test meals with 4L polyethylene glycol versus a clear liquid diet with 4L polyethylene glycol bowel preparation: a randomized trial. J Gastroenterol Hepatol. 2009 Jun;24(6):988-91. doi: 10.1111/j.1440-1746.2009.05860.x. PMID 19638081
- [Result] Rapier R, Houston C. A prospective study to assess the efficacy and patient tolerance of three bowel preparations for colonoscopy. Gastroenterol Nurs. 2006 Jul-Aug;29(4):305-8. doi: 10.1097/00001610-200607000-00007. PMID 16974167